CLINICAL TRIAL: NCT07210528
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of Emtricitabine and Descovy in Patients With Mild Cognitive Impairment.
Brief Title: Safety Of Nrtis for Alzheimer's Therapeutic Advancement in Singapore Study
Acronym: SONATAS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTi-EmtriDes-2022
Record Dates: First submitted 2025-07-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment (MCI); Alzheimer Dementia (AD)
Keywords: Reverse Transcriptase Inhibitors; Mild Cognitive Impairment (MCI); Descovy; Emtricitabine; Alzheimer's Disease (AD)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Emtricitabine; Racivir; emtricitabine tenofovir alafenamide; tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Descovy (Experimental): Equal numbers of male and female participants will be recruited in all arms. Descovy, Tablet, 200/25 mg, ct, Bottle, Britestock.
  Interventions: Drug: Descovy® (TAF/FTC)
- Placebo to Match Descovy (Placebo Comparator): Equal numbers of male and female participants will be recruited in all arms. Placebo to match Descovy. Tablets, Rectangular-Shaped, Debossed, Film-Coated Blue, 30ct per bottle.
  Interventions: Drug: Placebo to Match Emtricitabine 200mg/Tenofovir Alafenamide 25 mg.
- Emtricitabine (Emtriva) (Experimental): Equal numbers of male and female participants will be recruited in all arms. Emtriva, Capsule, 200 mg, 30 ct, Bottle, Britestock.
  Interventions: Drug: Emtricitabine (FTC)
- Placebo to match Emtricitabine (Emtriva) (Placebo Comparator): Equal numbers of male and female participants will be recruited in all arms. Placebo Capsules to Match Emtricitabine Capsules, 200 mg, White Opaque Body/Light Blue Opaque Cap with "GILEAD" and Gilead Logo on body, "200 mg" on cap printed in black, 30 ct per bottle.
  Interventions: Drug: Placebo Capsules to Match Emtricitabine Capsules, 200mg.

INTERVENTIONS:
Drug: Emtricitabine (FTC) — Capsule, 200mg FTC. White Opaque Body / Light Blue Opaque Cap with "GILEAD" and Gilead logo on body. "200 mg" on cap printed in black.
  Other Names: Emtriva
  Arms: Emtricitabine (Emtriva)
Drug: Descovy® (TAF/FTC) — Emtricitabine (FTC) 200 mg / Tenofovir Alafenamide (TAF) 25 mg. Tablets, Rectangular-Shaped, Debossed, Film-coated blue.
  Arms: Descovy
Drug: Placebo to Match Emtricitabine 200mg/Tenofovir Alafenamide 25 mg. — Placebo to Match Emtricitabine 200mg/Tenofovir Alafenamide 25mg. Tablets, Rectangular-Shaped, Debossed, Film-Coated Blue.
  Arms: Placebo to Match Descovy
Drug: Placebo Capsules to Match Emtricitabine Capsules, 200mg. — White Opaque Body/Light Blue Opaque Cap with "GILEAD" and Gilead logo on body, "200 mg" on cap printed in black.
  Arms: Placebo to match Emtricitabine (Emtriva)

SUMMARY:
Recent studies have identified an association between Alzheimer's Disease (AD) and an expansion of DNA content in the brain (prefrontal cortex). This additional DNA content appears to be derived from reverse transcriptase (RT) activity that incorporates genomic cDNAs (gencDNAs) into chromosomes, resulting in multiple copies of full length and shorter cDNAs involving many genes - including the causal AD gene amyloid precursor protein (APP). Accumulation of these APP gencDNAs is associated with AD.

This identifies RT as a promising therapeutic target for the attenuation of AD progression through existing reverse transcriptase inhibitors (RTi's) that have been widely used for treating HIV and hepatitis B. Since this class of drugs has been in the clinic for over 3 decades, there are significant data supporting their post-approval safety for long-term use. However, this has not been specifically addressed in the target population - patients with mild cognitive impairment (MCI), particularly women - who are underrepresented in HIV datasets.

This proposed Phase I safety trial will perform a Special Population Study in a cohort of MCI patients who may benefit from the intervention.

This study aims to (1) evaluate the safety and tolerability of standard dose FTC or Descovy for 3 months in MCI patients; (2) as secondary aims, collect preliminary data on clinical effects of standard dose FTC or Descovy compared to placebo for 3 months on cogntiive function in MCI patients; and (3) collect preliminary data on clinical effects of standard dose FTC or Descovy compared with placebo on AD-associated inflammatory markers.

Participants will be randomized into either Descovy or FTC arms in equal numbers, and receive either active drug or placebo. Participants will orally ingest 1 capsule or tablet (depending on drug arm) daily for the 3 month participation period.

The investigators hypothesise that MCI are not at increased risk of adverse effects due to administration of standard dose FTC or Descovy.

ELIGIBILITY:
Inclusion Criteria:

* MMSE score of 24 or above.
* CDR-GS of 0 or 0.5 (calculated by the QDRS)
* Diagnosed with MCI, determined by impairment in at least one domain of the neuropsychological test battery without significant dysfunction in activities of daily living OR MCI consistent with the NIA/AA diagnostic criteria.
* Does not have any medical condition (e.g. cardiac, respiratory, gastrointestinal, renal disease) which are not stably and adequately controlled, or which in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments.
* Willingness to provide blood sample and neuropsychological testing for the study.
* Ability for the patient to provide informed consent.

Exclusion Criteria:

* Patient who is receiving a prescription of acetylcholinesterase inhibitor (AChEI) and/or Memantine at screening or baseline.
* Patients with a history of HIV or HBV infection, or that test positive for HIV or HBV on screening.
* Pre-existing comorbidities such as Hepatits, cardiovascular disease, or renal insufficiency.
* History of Moderate to severe hepatic impairment indicated by screening AST or ALT > 3x the upper limit of normal (ULN) or total bilirubin > 2x ULN.
* Patients with severe renal impairment, or creatinine clearance ≤ 30 mL/min (calculated by Cockcroft-Gault formulae at screening).
* Co administration of nephrotoxic drugs.
* Current or previous RTi use within the last 2 years.
* Malignant neoplasm, and are undergoing active treatment.
* Participating in other interventional clinical trials during the course of the study.
* Documented history of lactic acidosis and severe hepatomegaly with steatosis.
* Documented history of osteoporosis.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related Adverse/Serious Adverse Events (AE/SAE) | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Number of participants with treatment-related AE/SAEs as assessed on the CTCAE Version 4.0. Incidence rate (n = x, and %), cause, and type of AE/SAE will be compared across the active drug and placebo groups.

SECONDARY OUTCOMES:
Change in circulating Beta-Amyloid 40 (Aβ40), Beta-Amyloid 42 (Aβ42) and Aβ-40: Aβ-42 ratio from baseline. | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Changes in plasma Aβ-40 and Aβ-42 levels; and Aβ40:Aβ42 ratio from baseline visit to week 12 visit, as assessed on Single Molecular Array (SIMOA). Units: pg/mL. No reference range is reported as significant variation exists across cohorts.
Change in Phospho-Tau217 (Ptau217) from baseline. | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Change in total plasma Ptau217 levels from baseline visit to week 12 visit, as assessed on Single Molecular Array (SIMOA). Units: pg/mL. No reference range is reported as significant variation exists across cohorts.
Change in Interleukin-6 (IL-6) levels from baseline. | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Change in serum IL-6 levels from baseline to week 12 visit, as assessed on Luminex Multiplex Analyser. Units: pg/mL. No reference range is reported as significant variation exists across cohorts.
Change in Interleukin-8 (IL-8) levels from baseline. | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Change in serum IL-8 levels from baseline to week 12 visit, as assessed on Luminex Multiplex Analyser. Units: pg/mL. No reference range is reported as significant variation exists across cohorts.
Change in Tumor Necrosis Factor-alpha (TNFα) levels from baseline. | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Change in serum TNFα levels from baseline to week 12 visit, as assessed on Luminex Multiplex Analyser. Units: pg/mL. No reference range is reported as significant variation exists across cohorts.
Change in Mini Mental State Exam scores (MMSE). | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Change in MMSE total scores from baseline visit to week 12 visit, to assess changes in cognitive function. Scores range from 0 - 30, with higher scores indicating better cognitive function.
Change in Quick Dementia Rating Scores (QDRS) from baseline. | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Change in QDRS total scores from baseline visit to week 12 visit, to assess changes in cognitive function. Scores range from 0 - 30, with higher scores indicating greater cognitive and functional impairment.
Change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) scores from baseline. | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Change in RBANS total and index scores from baseline to week 12 visit to assess changes in cognitive function. The battery consists of 5 indexes: 1) Immediate Memory, 2) Visuospatial/Constructional, 3) Language, 4) Attention, and 5) Delayed Memory and 12 subtests which are indexed and scored according to standardized RBANS criteria - adjusting for age and education):
  Immediate Memory: List Learning, Story Memory; Visuospatial/Constructional: Figure Copy, Line Orientation; Language: Picture Naming, Semantic Fluency; Attention: Digit Span, Coding; Delayed Memory: List Recall, List Recognition, Story Recall, Figure Recall.
  Raw scores of all 12 subtests will be converted to age- and education-adjusted scaled scores before calculating an index score for each domain. Sum of index scores will then be converted to a Total Scale score. Scaled scores range from 40 - 160, with higher scores indicating higher overall cognitive function.
Change in Colour Trials Test (CTT) scores from baseline. | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Change in CTT (Trial 1 & 2) completion times from baseline to week 12 visit, to assess changes in attention and sequencing. Units: Time-to-completion (seconds) for each Trial. A range of time-to-completion of 3-8 minutes is reported in the CTT manual, with longer completion times indicative of impaired attention and sequencing.
Change in Activities of Daily Living (ADL) scores from baseline. | From enrollment to the end of treatment at 12 weeks (measured from participant's baseline visit).
  Change in Independent ADL scores from baseline to week 12 visit, as assessed on the Activities of Daily Living Preventative Instrument (ADCS-ADL-PI) - comprising 15 ADL and 5 physical function questions covering complex activities typically conducted by most during independent living (e.g. handling money, shopping, remembering plans and appointments).
  ADLs are scored on a 5-point Likert scale. Total scores range from 0 - 45, with higher scores indicating less functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chen, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Sensitive health information will be collected as part of this study. Only de-indentified data will be used for study purposes.